CLINICAL TRIAL: NCT05982301
Title: PD-1 Antibody Sintilimab Combined With Modified FLOT Regimen in the Treatment of Metastatic Gastric Cancer: a Phase II Clinical Study
Brief Title: Sintilimab Combined With Modified FLOT Regimen in the Treatment of Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, Director, Head of Gastrointestinal Oncology, Principal Investigator, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-PFMG
Record Dates: First submitted 2023-05-19; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Gastric Cancer; Chemotherapy Effect; Immune Checkpoint Inhibitor
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nab-POF (Experimental): Sintilimab 200mg d1 ivgtt+paclitaxel-albumin 125mg/m2 d1 ivgtt+oxaliplatin 85mg/m2 d1 ivgtt+5-FU 2.4g/m2 civ46h, q2w.
  Interventions: Drug: Sintilimab, paclitaxel-albumin, oxaliplatin, 5-FU

INTERVENTIONS:
Drug: Sintilimab, paclitaxel-albumin, oxaliplatin, 5-FU — The study has only one arm. Sintilimab 200mg d1 ivgtt+paclitaxel-albumin 125mg/m2 d1 ivgtt+oxaliplatin 85mg/m2 d1 ivgtt+5-FU 2.4g/m2 civ46h, q2w.
  Other Names: Sintilimab+mFLOT

SUMMARY:
This is a prospective, one-arm, single-center phase II study. The objective was to evaluate the efficacy and safety of domestic PD-1 antibody Sintilimab combined with modified FLOT regimen in the treatment of metastatic gastric cancer. To compare the time of maintenance of treatment after induction of chemotherapy with sintilimab combined with modified FLOT regimen until the reapplication of induction regimen with or without the combination of sintilimab, and the time of secondary progression after signing informed consent until the reapplication of induction regimen with or without the combination of sintilimab.

DETAILED DESCRIPTION:
This study set up two cohorts, Cohort A: patients with HER2-negative advanced gastric cancer, and planned to enroll 87 patients with initially treated advanced gastric cancer. Thirty patients with ORR of more than 70% were enrolled in the first stage and then further enrolled. Cohort B: advanced gastric cancer patients with HER2 positive initial treatment, the number of enrolled is not specified. Patients with initially treated advanced gastric cancer who meet the inclusion criteria will be enrolled in this study to receive Sintilimab combined with mFLOT regimen. Trastuzumab was given to Cohort B. The results were repeated every 2 weeks and evaluated every 6 weeks. The examination methods were consistent with those at baseline. Patients without disease progression were treated for a maximum of 6 cycles, then switched to oral capecitabine monotherapy combined with the sintilimab until disease progression, intolerable adverse reactions, patient death, or withdrawal of informed consent. If intolerability toxicity of albumin paclitaxel or oxaliplatin occurs within 6 cycles, maintenance is advanced to sintilimab combined with capecitabine monotherapy. Patients were randomly assigned to Cohort A1 and Cohort A2 after maintaining treatment progress. Cohort A1: Cohort 1 combined with mFLOT; Cohort A2: mFLOT program Therapy. The regimen was repeated every 2 weeks and tumor efficacy was evaluated every 3 treatment cycles. Patients without disease progression were treated for a maximum of 6 cycles before being switched to monotherapy S-1 oral with or without sintilimab until disease progression, intolerable adverse reactions, patient death, or withdrawal of informed consent. The treatment should start within 1 week after the signing of informed consent, and the time from the signing of informed consent to the first progress should be PFS1; The time from the signing of informed consent to the progress of induction program back to the second progress is PFS2. In this study, peripheral blood and tissue samples of patients will be collected to analyze the correlation between biomarkers (such as Micro-RNA, cytokine expression levels, etc.) and efficacy and prognosis. The expected time of enrollment was 48 months, and the patients were observed clinically until disease progression and death. (PFS2 equals PFS1 if the induction regimen is applied again after the first disease progression and the first efficacy evaluation is the disease progression)

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years and men or women
2. With histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction, local lesions that cannot be radically resected, or metastatic gastric cancer
3. For treatment-naïve patients, or postoperative recurrence at least 6 months from the last adjuvant chemotherapy
4. With Eastern Cooperative Oncology Group (ECOG) PS of 0-1
5. With a life expectancy of more than 3 months
6. Who obtain the following laboratory test data within 7 days (including the seventh day) prior to the study screening: neutrophil count of ≥1.5 × 10^9/L, platelet count of ≥100 × 10^9/L, hemoglobin level of ≥90 g/L, serum total bilirubin of ≤1.25 the upper limit of normal (ULN); ALT and AST levels of ≤2.5 × ULN (≤5 × ULN for patients with liver metastasis); serum creatinine level of ≤1.0 × ULN and creatinine clearance of ≥50 ml/min; International Normalized ratio (INR) or prothrombin time (PT) ≤1.5 ULN; If the subject is receiving anticoagulant therapy, PT should be within the prescribed anticoagulant range.
7. With at least one extragastric measurable lesion (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria)
8. Patients (or their legal representative/guardian) must sign an informed consent form indicating that they understand the purpose of the study, understand the procedures necessary for the study, and are willing to participate in the study.

Exclusion Criteria:

1. Patients with history of other types of cancer in the last 3 years, except for cured cervical cancer or cutaneous basal cell carcinoma.
2. Patients with symptomatic brain or leptomeningeal metastases (unless the patient has been treated for >2 months) who has a negative imaging result within 4 weeks before participating in the study and is stable disease at study entry.
3. Patients with clinically significant gastrointestinal obstruction, gastrointestinal bleeding (defecate occult blood + + + and above) or perforation.
4. Patients who have received PD-1, PD-L1 or PD- L2, CD137, CTLA-4 antibody therapy, or any other T cells stimulate or total checkpoint pathways for specific target antibody or drugs.
5. Patients with active, or have a history and possible recurrence of autoimmune disease of the subjects (such as: Systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.), or those at high risk (such as those who have received an organ transplant requiring immunosuppressive therapy). However, patients with vitiligo, psoriasis, alopecia, or Grave's disease who did not require systemic treatment within the last 2 years, or patients with hypothyroidism who required only thyroid hormone replacement therapy, and patients with type 1 diabetes who required only insulin replacement therapy could be enrolled.
6. Patients now with interstitial lung disease or pneumonia, pulmonary fibrosis, acute lung diseases, radiation pneumonia.
7. Patients who received any investigational drugs or antitumor drugs within 4 weeks prior to enrollment.
8. Patients who received immunosuppressive drugs within 4 weeks, which does not include nasal, inhalation or other routes of topical corticosteroids or physiological doses of systemic corticosteroids (i.e., not exceeding 10 mg/ day of prednisone or equivalent doses of other corticosteroids), or short-term (not exceeding 7 days) use of corticosteroids for the prevention or treatment of non-autoimmune allergic diseases.
9. Patients who received the live attenuated vaccine within 4 weeks before the first dose of study treatment. Note: Inactivated virus vaccines for injectable seasonal influenza are permitted for up to 4 weeks prior to initial administration; But live attenuated influenza vaccines are not allowed;
10. Patients who received major surgery within 4 weeks before the first dose of study treatment(open chest, craniotomy or laparotomy) or expected during the research and treatment need to accept major surgery not associated with this study.
11. Patients who infected with human immunodeficiency virus (HIV) disease (HIV antibody positive), or with other acquired, congenital immunodeficiency disease, or has a history of organ transplantation, or stem cell transplantation.
12. Patients who have chronic active hepatitis B or active active hepatitis C. Hepatitis B virus carriers, stable after drug treatment of hepatitis B (DNA drop degree is not higher than 200 iu/mL or copy number < 1000 copies/mL) and has cured patients with hepatitis c (HCV RNA test negative) into the group.
13. Patients with known active tuberculosis.
14. Patients with severe infections before 4 weeks of fisrt dose of treatment, active infection which needs oral or intravenous antibiotic therapy before 4 weeks of fisrt dose of treatment.
15. Patients with symptomatic congestive heart failure (New York heart association grade II - IV) or symptomatic or poorly controlled arrhythmia.
16. Patiemts with uncontrolled arterial blood pressure with specification treatment (systolic blood pressure of greater than 160mmHg or diastolic blood pressure of greater than 100 mmHg).
17. Patients who had any arterial thromboembolic events, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack within 6 months before the screening.
18. Patinets with deep vein thrombosis, pulmonary embolism, or any other serious history of thromboembolism within 3 months (implantable venous infusion port source sex or catheter thrombosis, or superficial venous thrombosis were not regarded as a "severe" thromboembolism).
19. Patients who have a history of neurological or psychiatric disorders, such as memory, epilepsy, dementia, compliance, or the peripheral nervous system disorder.
20. alcohol dependence or 1-year history of drug or drug abuse.
21. Pregnancy or lactation women; Those who are fertile but do not take adequate contraceptive measures;
22. may lead to the following results of other acute or chronic diseases, mental illness or abnormal laboratory values: participated in or study drug dosage associated with an increased risk, or interfere with the interpretation of results, and according to the researcher's judgment does not conform the patient to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free survival 2, PFS2 | From date of informed consent to time of secondary progression, assessed up to 60 months
  From date of informed consent to time of secondary progression

SECONDARY OUTCOMES:
Overall survival, OS | the period from the date of randomization to the date of death from any cause, assessed up to 60 months
  the period from the date of randomization to the date of death from any cause.
Objective response rate | Baseline, Every 6 weeks during the procedure, up to 1 year. After 1 year, every 3 months.
  the proportion of patients whose tumor dcrease to a certain size and remained for a certain period of time, including those with complete response(CR) and partial response (PR).
Progression-Free survival 1, PFS1 | From date of informed consent to time of first progression, assessed up to 60 months.
  From date of informed consent to time of first progression
After Effects | Baseline, Every cycle of treatment, until disease progression or death, whichever come first.
  CTC AE Version 5.0 will be used to evaluate the clinical safety of the treatment in the study.

CONTACTS AND LOCATIONS:
Overall Officials: WeiJian Guo, M.D.,Ph.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to share IPD after the publication of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We plan to share IPD after the publication of the study.
Access Criteria: Data sharing requires approval from the principal investigator.